CLINICAL TRIAL: NCT04380402
Title: Prospective Randomized Open-label Trial of Atorvastatin as Adjunctive Treatment of COVID-19
Brief Title: Atorvastatin as Adjunctive Therapy in COVID-19
Acronym: STATCO19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Auburn Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MountAuburn
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 40 mg
  Interventions: Drug: Atorvastatin
- Control (No Intervention): Standard care

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40 mg tablet
  Other Names: atorvastatin calcium
  Arms: Treatment

SUMMARY:
Objective: To assess whether adjunctive therapy of COVID-19 infection with atorvastatin reduces the deterioration in hospitalized patients and improves clinical outcome.

DETAILED DESCRIPTION:
COVID-19 is caused by SARS-CoV-2, a β-coronavirus that binds to the zinc peptidase angiotensin-converting enzyme 2 (ACE2). No drug is licensed to treat COVID-19, but adjunctive pharmacologic interventions have been proposed for their immunomodulatory effects, including statins. About 5% of cases are considered critical, with severe respiratory failure as well as myocarditis, and thromboses, and are associated with high fatality rate. Statins affect endothelial dysfunction and have anti-inflammatory and immunomodulatory effects.

This prospective, randomized, open-label trial of atorvastatin as adjunctive treatment of COVID-19 in hospitalized patients aims to study:

1. Will atorvastatin reduce progression to severe or critical COVID-19 disease and death compared to standard care?
2. Will atorvastatin lead to improved clinical outcome of COVID-19 disease at 30 days compared to standard care?

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-85 years, admitted with suspected COVID-19 disease based on clinical criteria (typical upper respiratory symptoms, e.g. runny nose, sore throat, dry cough, associated with COVID-19 infection).

Exclusion Criteria:

* already on chronic statin therapy, known hypersensitivity or adverse events to statins, negative nasopharyngeal (NP) swab for SARS-CoV-2, pregnancy and lactation, need for ICU admission, ALT or AST >2X upper limit of normal; CPK > 5x upper limit of normal; and creatinine clearance <50%, chronic treatment with colchicine, cyclosporin, digoxin, fusidic acid, azole antifungals, niacin.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that progress to severe or critical requiring ICU admission and/or emergency salvage therapy, or death | 30 days
  Proportion of patients in each arm that progress to severe or critical requiring ICU admission and/or emergency salvage therapy, or death, as described by WHO Ordinal Scale for Clinical Improvement scores 5-8 with higher being worse.

SECONDARY OUTCOMES:
Overall score of patients in each arm on Day 7 based on WHO Ordinal Scale for Clinical Improvement | 7 days
  Description of clinical status of patients in each arm based on WHO Ordinal Scale of Clinical Improvement on Day 7, scores 1-8 with higher being worse.
Overall score of patients in each arm on Day 30 based on WHO Ordinal Scale for Clinical Improvement | 30 days
  Description of clinical status of patients in each arm based on WHO Ordinal Scale of Clinical Improvement on Day 30, scores 1-8 with higher being worse.
Proportions of patients in each arm who test negative for SARS-CoV-2 on Day 7 | 7 days
  Proportions of patients in each arm who are tested on Day 7 and have negative PCR

CONTACTS AND LOCATIONS:
Overall Officials: Lin H Chen, MD, Principal Investigator — Mount Auburn Hospital
Locations (1):
- Mount Auburn Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Parihar SP, Guler R, Brombacher F. Statins: a viable candidate for host-directed therapy against infectious diseases. Nat Rev Immunol. 2019 Feb;19(2):104-117. doi: 10.1038/s41577-018-0094-3. PMID 30487528
- [Background] Vandermeer ML, Thomas AR, Kamimoto L, Reingold A, Gershman K, Meek J, Farley MM, Ryan P, Lynfield R, Baumbach J, Schaffner W, Bennett N, Zansky S. Association between use of statins and mortality among patients hospitalized with laboratory-confirmed influenza virus infections: a multistate study. J Infect Dis. 2012 Jan 1;205(1):13-9. doi: 10.1093/infdis/jir695. Epub 2011 Dec 13. PMID 22170954
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Fedson DS, Opal SM, Rordam OM. Hiding in Plain Sight: an Approach to Treating Patients with Severe COVID-19 Infection. mBio. 2020 Mar 20;11(2):e00398-20. doi: 10.1128/mBio.00398-20. PMID 32198163
- See also: Statin therapy in acute influenza — https://clinicaltrials.gov/ct2/show/results/NCT02056340?view=results